CLINICAL TRIAL: NCT01208753
Title: Double Blind Placebo Controlled Dose Ranging Study for the Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Oral Doses of GLPG0555 in Healthy Subjects.
Brief Title: Pharmacokinetics/Pharmacodynamics (PK/PD) of Multiple Oral Doses of GLPG0555 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Senior Vice President Development, Galapagos NV
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLPG0555-CL-102; 2010-018570-20 (EudraCT Number)
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aqueous formulations for formulation selection (Experimental): 50 mg once daily for 3 days of two different aqueous suspensions, with four day wash-out between formulation
  Interventions: Drug: GLPG0555
- GLPG0555 ascending doses (Experimental): multiple ascending doses for 13 days, ranging from 100 mg once daily upto a maximum to be determined during escalation (given as once or twice daily)
  Interventions: Drug: GLPG0555 aqueous
- 3 (Placebo Comparator): once or twice daily for 13 days, matching the scheme of the multiple ascending dose.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GLPG0555 — two different aqueous formulations
  Arms: Aqueous formulations for formulation selection
Drug: GLPG0555 aqueous — multiple dose, aqueous formulation, 13 days, 100 mg/day once daily, maximum dose to be determined
  Arms: GLPG0555 ascending doses
Drug: placebo — multiple dose, aqueous formulation, 13 days days, matching ascending dose schedule
  Arms: 3

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple ascending oral doses (MAD) of GLPG0555 given to healthy subjects for 13 days compared to placebo, and to evaluate the relative bioavailability and pharmacokinetics (PK) of two different aqueous suspensions of GLPG0555 administered for 3 days. Finally, it is aimed to characterize PK and pharmacodynamics (PD) of GLPG0555 after multiple oral administrations.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m², inclusive.

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple dosing | Daily during treatment, up to 10 days postdose

SECONDARY OUTCOMES:
Pharmacokinetics of repeated doses | 24 hours postdose
Pharmacodynamics (PD) of GLPG0555 after repeated oral administration | up to 10 days postdose
The relative bioavailability and pharmacokinetics (PK) of two different aqueous suspensions administered for three days | up to 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Gerben van 't Klooster, PhD, Study Director — Galapagos NV; Wouter Haazen, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium